CLINICAL TRIAL: NCT02469584
Title: Continuous Small Stitch Technique for Anterior Colporrhaphy: a Pilot Study
Brief Title: Small Stitch Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Halpern Ksenia, Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1236/2014
Record Dates: First submitted 2015-06-05; First posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Anterior Vaginal Wall Prolapse
Keywords: prolapse; anterior colporrhaphy
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): symptomatic cystocele described as Points Aa or Ba >= 0 according to the International Continence Society pelvic organ prolapse quantification system (POP-Q). The changes in POPQ score preoperatively and three months after the anterior colporrhaphy with the new small stitch technic will be analyzed.
  Interventions: Procedure: small stitch anterior colporrhaphy

INTERVENTIONS:
Procedure: small stitch anterior colporrhaphy — A midline plication will be performed with continuous delayed absorbable sutures (3-0 polydioxanone) and the distance between the sutures will be 0.5 cm.

SUMMARY:
A descent of the anterior vaginal wall is the most common form of female pelvic organ prolapse (POP). Although anterior colporrhaphy (AC) is accepted worldwide as a "standard procedure", its exact steps are not well standardized.

We developed a small stitch anterior colporrhaphy (SSTAC) in an effort to increase the strength and durability of AC

Objectives

The aim of this pilot study is to demonstrate the feasibility and complication rate of the SSTAC and to assess the anatomical and functional outcomes after this method of cystocele repair.

DETAILED DESCRIPTION:
A prospective case series evaluation of SSTAC following the recommendations of IDEAL-Collaboration (www.ideal-collaboration.net) will be performed. The newly developed procedure will be tested in a group of 10 patients, who equals stage 2a in the development and innovation of surgical innovations. In this stage safety and technical success is the main outcome. As technical modifications may be common during stage 2a and their nature and timing should be meticulously recorded, the videotaping during all surgical procedures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* women older than 18 years of age
* Able to read, understand and sign informed consent
* symptomatic cystocele described as Points Aa or Ba >= 0 according to the International Continence Society pelvic organ prolapse quantification system (POP-Q)

Exclusion Criteria:

* previous urogynecological operation
* gynecologic malignancy
* planned concomitant incontinence operation
* other contraindications for surgery
* pregnancy
* systemic glucocorticoid treatment
* contraindication for the surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
the most distal point of the anterior vaginal wall- postoperative anterior vaginal support described as Point Ba (POP-Q score) | 4-6 weeks, 3 months
  The changes in POPQ score preoperatively and three months after the anterior colporrhaphy with the new small stitch technic will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Engelbert Hanzal, Dr, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria, Austria